CLINICAL TRIAL: NCT02124031
Title: Mexican Initiative of Patients With Osteoarthritis and Rheumatoid Arthritis
Brief Title: Mexican Initiative of Patients With Osteoarthritis and Rheumatoid Arthritis (IMPACTAR)
Acronym: IMPACTAR
Status: Completed | Type: Observational
Sponsor: Iniciativa Mexicana de Pacientes con Osteoartritis y Artritis Reumatoide (Other)
Collaborators: Sanofi (Industry); Webmedica (Unknown)
Responsible Party: Sponsor
Other Study IDs: IMPACTAR
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Physical Disability; Joint Function Disorder; Axis IV Problems Economic; Compliance Behavior; Complications; Arthroplasty
Keywords: Osteoarthritis; Rheumatoid Arthritis; Disability; Joint function
MeSH Terms: conditions — Patient Compliance; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate quality of life, degree of disability, treatment patterns and economic impact of hand and knee Osteoarthritis and Rheumatoid Arthritis in Mexico.

DETAILED DESCRIPTION:
The osteoarthritis (OA) is a chronic and degenerative disease of multifactorial etiology, characterized by the gradual loss of articular cartilage. It is a question of one of the most common rheumatic disorders in the population, is the most habitual reason of pain and disability in the major adults and the first reason of surgeries of articular replacement. In Mexico, in a study of national area, the prevalence of locomotives manifestations was 26 %, with predominance in the women. Nowadays criteria exist for the classification of the OA, based on epidemiological studies, for the knee, the hip and the hand. Basically they have been established to homogenize studies of clinical epidemiological type. In other hand, the Rheumatoid Arthritis (RA) is an inflammatory, chronic, systemic disease that has more prominent manifestations in the diarthrodial joints. The disease have a wide range of characteristics, from the progressively chronic disease with variable degrees of destruction to articulate up to the extra-articular manifestations clinically evident. Demographically, the RA is the most common form of inflammatory arthritis and affects approximately 0.5 to 1 % of the world population, with an economic impact comparable with arterial coronary disease. The National Institute of Geographical Statistics (INEGI) thinks that in Mexico the population of major adults will double in the next decades, for what the impact of these rheumatic disorders will be serious and will turn into a problem of public health.

Based in the previous information, the Mexican Initiative of Patients with OA and RA (IMPACTAR), will on patient interview to increase the knowledge regarding the number of affected adults and the current treatment strategies.

This will be the first Mexican Registry related with Osteoarticular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years with diagnosis of OA or RA according to the criteria of the American College of Rheumatology (ACR).

Exclusion Criteria:

* Patients with precedents of fractures; carrying patients of chronic diseases who limit them in the functional capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Registry will include male and female patients older than 18 years with knee and/or hand OA and/or RA diagnosis according with the American College of Rheumatology criteria. It will include consecutive outpatients that are treated in any of the participant specialties of the study (orthopedics, rheumatology, internal medicine, rehabilitation medicine).
Sampling Method: Probability Sample
Enrollment: 10241 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | Previous six months
  For evaluate the impact in quality of life we will use the EUROQoL score

SECONDARY OUTCOMES:
Articular function | Previous six months
  For evaluate the impact for articular function we will use the MDHAQ score, m-SACRAH score (hand) and WOMAC score (knee)

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Espinosa, M. D., Principal Investigator — National Institute of Rehabilitation